CLINICAL TRIAL: NCT01956929
Title: Metformin's Effect on Glucagon-induced Endogenous Glucose Production, Protein Metabolism and Resting Energy Expenditure in Insulin Resistant Individuals.
Brief Title: Metformin's Effect on Glucagon-induced Glucose Production and Protein Metabolism.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-004966
Record Dates: First submitted 2013-09-23; First posted 2013-10-08 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance; Prediabetic State
Keywords: Insulin Resistance; Prediabetic State; Metformin
MeSH Terms: conditions — Insulin Resistance; Prediabetic State | interventions — Metformin; Lactulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): 2 weeks of Metformin use. First week 1000mg/day, Second week Max dose of 2000 mg/day.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 2 weeks of Placebo (lactulose pills)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg daily for one week, then 2000 mg daily for the second week. 4 week washout period, then crossover to placebo.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Placebo tablets for 2 weeks, then 4 weeks of washout period, then crossover to metformin.
  Other Names: Lactulose
  Arms: Placebo

SUMMARY:
This study is being done to understand metformin's mechanisms of action regarding glucose production, protein metabolism, and mitochondrial function.

DETAILED DESCRIPTION:
It is believed that Metformin antagonizes the action of glucagon through different pathways. In mice, Metformin leads to inhibition of adenylate cyclase, reduction of levels of cyclic AMP and protein kinase A (PKA) activity, therefore blocking glucagon-dependent glucose output form hepatocytes. Glucagon plays an important role in the increased catabolic state seen in insulin deficiency. Hyperglucagonaemia states have been shown to accelerate proteolysis and leucine oxidation in insulin-deficient humans. Patients with insulin resistance and increased levels of glucagon have an increased in energy expenditure which may contribute to the catabolic state associated with this condition. We hypothesized that treatment with Metformin for 2 weeks will significantly inhibit glucagon-induced endogenous glucose production in insulin resistant individuals. We also hypothesized that glucagon-induced alterations in whole body protein metabolism and the increases in O2 consumption associated with hyperglucagonaemia states will be significantly inhibited by Metformin in these individuals. This would open the door for the development of other antidiabetic drugs with antagonism of glucagon as their principal mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* 35-65 years of age
* Fasting blood glucose >100 mg/dl
* BMI 27-36 kg/m2
* Waist Circumference: Men ≥ 104 cm; women ≥ 88 cm
* If previously on anti-diabetic medication, should be off for at least 1 month

Exclusion Criteria:

* Active use of hypoglycemic agents (< 1 month)
* Renal failure, creatinine ≥ 1.5 mg/dL in men or ≥ 1.4 mg/dL in women
* Alanine aminotransferase levels exceed 135 IU/L or aspartate aminotransferase levels exceed 129 IU/L (3 x the upper limit of normal)
* Congestive Heart Failure (EF < 40 %)
* Active coronary artery disease
* Recent (less than 6 weeks) or planned imaging study requiring IV contrast
* Participation in structured exercise (> 2 hr per week)
* Recent change in dietary habits or weight
* Tobacco use
* Use of systemic glucocorticoids
* Anti-coagulant therapy (warfarin/heparin)
* Pregnancy or breastfeeding
* Alcohol consumption greater than 2 drinks/day
* Uncontrolled Hypothyroidism, abnormal thyroid stimulating hormone levels
* Metformin Allergy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Glucagon-induced endogenous glucose production. | Measured at week 0, 2, 4, 6 and 8
  To assess the effect of Metformin on glucose metabolism, at baseline and during a period of hyperglucagonemia, endogenous glucose production will be measured using a stable isotope tracer during the application of a somatostatin-based pancreatic clamp. Participants will be assessed before and following two weeks of consuming either metformin or placebo.

SECONDARY OUTCOMES:
Change in glucagon-induced alterations in whole body protein metabolism and resting energy expenditure. | Measured at week 0, 2, 4, 6 and 8
  Alterations in whole body protein metabolism will be measured by using leucine as a tracer that measures leucine flux, and leucine transamination and oxidation as measures of leucine catabolism. Whole body oxygen consumption will be assessed by open circuit indirect calorimetry with a ventilated hood system. Skeletal muscle biopsies will be obtained at baseline and four hours after a high fat, high glycemic meal. Mitochondria will be isolated from the muscle samples to assess mitochondrial oxygen consumption and hydrogen peroxide emissions using high-resolution respirometry and spectrofluorometry, respectively. In addition, we will measure skeletal muscle intracellular AMP-activated protein kinase activity.

CONTACTS AND LOCATIONS:
Overall Officials: K Nair, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States